CLINICAL TRIAL: NCT02698449
Title: Cognitive Rehabilitation Combined to Transcranial Direct Current Stimulation Following Traumatic Brain Injury: Functional Magnetic Resonance Imaging Study
Brief Title: Neurorehabilitation After Traumatic Brain Injury: Functional Magnetic Resonance Imaging Study
Acronym: RemCog-TC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/14/7328
Record Dates: First submitted 2016-02-18; First posted 2016-03-03 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cognitive rehabilitation + transcranial stimulation (Experimental): specific cognitive rehabilitation combined to transcranial direct current stimulation
  Interventions: Procedure: transcranial direct current stimulation; Procedure: Specific cognitive rehabilitation; Radiation: functional Magnetic Resonance Imaging n-back task
- cognitive rehabilitation + stimulation sham (Experimental): specific cognitive rehabilitation combined to transcranial direct current stimulation sham
  Interventions: Procedure: Specific cognitive rehabilitation; Procedure: transcranial direct current stimulation sham; Radiation: functional Magnetic Resonance Imaging n-back task
- placebo rehab + transcranial stimulation (Experimental): nonspecific cognitive rehabilitation (placebo rehab) combined to transcranial direct current stimulation
  Interventions: Procedure: transcranial direct current stimulation; Procedure: Nonspecific cognitive rehabilitation; Radiation: functional Magnetic Resonance Imaging n-back task
- placebo rehab + stimulation sham (Experimental): nonspecific cognitive rehabilitation (placebo rehab) combined to transcranial direct current stimulation sham
  Interventions: Procedure: Nonspecific cognitive rehabilitation; Procedure: transcranial direct current stimulation sham; Radiation: functional Magnetic Resonance Imaging n-back task

INTERVENTIONS:
Procedure: transcranial direct current stimulation — intensity provided will be 2 milliampere during 20 minutes using 2 electrodes (7x5cm). Anode electrode will be located on the right prefrontal dorsolateral area; cathode electrode will be located on the left supraorbital area.
  Arms: cognitive rehabilitation + transcranial stimulation; placebo rehab + transcranial stimulation
Procedure: Specific cognitive rehabilitation — Specific cognitive rehabilitation will be personalized regarding the cognitive complaint and will include a training part and an ecological part.
  Arms: cognitive rehabilitation + stimulation sham; cognitive rehabilitation + transcranial stimulation
Procedure: Nonspecific cognitive rehabilitation — Nonspecific cognitive rehabilitation will be focused on representation of body in space.
  Arms: placebo rehab + stimulation sham; placebo rehab + transcranial stimulation
Procedure: transcranial direct current stimulation sham — the same operation that transcranial direct current stimulating but it is a sham surgery
  Arms: cognitive rehabilitation + stimulation sham; placebo rehab + stimulation sham
Radiation: functional Magnetic Resonance Imaging n-back task — the n-back cognitive task was developed : 3 runs will be provided (0-back, 1-back and 2-back), each will be composed of 8 activation blocks and 8 resting blocks alternatively presented.

SUMMARY:
The current study aims to better understand cerebral plasticity mechanisms to optimize non-pharmacological rehabilitation approaches for patients with traumatic brain injury.

DETAILED DESCRIPTION:
Cognitive impairment following moderate to severe traumatic brain injury are usual. To date, cognitive rehabilitation effects on cerebral plasticity and quality of life remain unproven essentially because of methodological biases. Transcranial Direct Current Stimulation is an innovative technique of noninvasive brain stimulation that showed efficacy in literature. The current study want to better understand cerebral plasticity mechanisms to optimize non-pharmacological rehabilitation approaches for patients with traumatic brain injury. The aim in the present study is to assess the effect of rehabilitation combined with Transcranial Direct Current Stimulation provided to traumatic brain injury patients with cognitive impairment on cerebral plasticity using functional magnetic resonance imaging. Effects of rehabilitation and Transcranial Direct Current Stimulation will be observed on functional magnetic resonance imaging activation maps acquired. Relationship between attentional outcomes measured in the neuropsychological assessment and activation extend will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe traumatic brain injury
* more than 3 months since the onset
* Attentional disorders (PASAT test (score ≤ centile 10) and/or CANTAB test (≤ -2 standard deviation)
* Women having contraceptive treatment (for the magnetic resonance imaging exam)

Exclusion Criteria:

* inability to undergo magnetic resonance imaging scan
* No attentional impairment (PASAT ≥ centile10)
* Severe depression
* Neurological disease
* Major cognitive impairment (aphasia, neglect)
* Drugs addiction
* Pregnant women and women having no contraceptive treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-01-24 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
intergroup difference on cerebral map activation in functional magnetic resonance imaging (N-back task). | 12 weeks

SECONDARY OUTCOMES:
Intergroup differences in resting activation maps. | 12 weeks
Intergroup differences in diffusion measures | 12 weeks
Intergroup differences in neuropsychological score | 12 weeks
Correlation between activation extend and attentional outcomes | 12 weeks
Intergroup differences in polymorphisms | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie Pariente, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No